CLINICAL TRIAL: NCT00151385
Title: A Multicenter Study to Describe the Immunogenic Epitope(s) of Factor VIII in Previously Treated Patients With Congenital Hemophilia A Who Develop De Novo Factor VIII Inhibitors While Receiving Factor VIII Infusion Therapy.
Brief Title: Study Evaluating Inhibitor Specificity in Hemophilia A
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3082A-101342
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: single blood draw

SUMMARY:
This investigation will utilize a systematic determination of anti-FVIII antibody specificity in PTPs (> 50 ED) with hemophilia A who have developed inhibitors in response to treatment with any FVIII product(s). A group of patients with hemophilia A, who have no evidence of current or prior FVIII inhibitor will be included for comparison. The objective of this study is to describe the patterns of antibodies and associated epitopes in the study population.

ELIGIBILITY:
Inclusion Criteria:

· Patients with moderate or severe congenital hemophilia A, a current FVIII inhibitor, who have taken at least two different FVIII products during their lifetime.

Exclusion Criteria:

* Patients who have had an inhibitor prior to their current inhibitor.
* Patients with immune disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-11; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Description of the patterns of antibodies and associated epitopes in a subset of
previously treated patients with hemophilia A.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trail Manager, Principal Investigator — For Italy, decresg@wyeth.com; Trial Manager, Principal Investigator — For Spain, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For UK, ukmedinfo@wyeth.com; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Germany, MedInfoDEU@wyeth.com
Locations (23):
- United States (7):
  - Atlanta, Georgia
  - Detroit, Michigan
  - New Hyde Park, New York
  - New York, New York
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - San Antonio, Texas
- Belgium (2):
  - Brussels
  - Leuven
- France (3):
  - La Bouëxière
  - Le Kremlin-Bicêtre
  - Lyon
- Germany (5):
  - Berlin
  - Bonn
  - Bremen
  - München
  - Münster
- Italy (2):
  - Florence
  - Milan
- Spain (2):
  - Madrid
  - Valencia
- United Kingdom (2):
  - London
  - Manchester